CLINICAL TRIAL: NCT06749444
Title: Cognitive Behavioral Therapy for Sleep and Circadian Disturbances (CBT-I) in Treatment-Resistant Schizophrenia
Acronym: COSTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jimmi Nielsen (Other)
Responsible Party: Sponsor-Investigator, Jimmi Nielsen, Professor, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24002249; 10.46540/3166-00056B (Other Grant/Funding Number: DFF: Independent Research Fund Denmark)
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-08

CONDITIONS: Treatment-refractory Schizophrenia; Treatment-resistant Schizophrenia
Keywords: Cognitive; CBT; Therapy; Insomnia; polysomnography
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Sleep laboratory employees
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy for insomnia (Experimental): 8-10 sessions CBT-I tailored for insomnia symptoms
  Interventions: Other: CBT-I
- Cognitive Behavioral Therapy (Active Comparator): 8-10 sessions CBT tailored for general psychopathology
  Interventions: Other: CBT

INTERVENTIONS:
Other: CBT-I — Cognitive therapy tailored for insomnia symptoms.
  Other Names: Cognitive behavioral therapy for insomnia
  Arms: Cognitive Behavioral Therapy for insomnia
Other: CBT — Cognitive behavioral therapy for general psychopathology
  Other Names: Cognitive behavioral therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
Using a randomized controlled design, the project aims to test if cognitive behavioral therapy interventions specifically targeting sleep disorders can significantly lessen the burden of the disrupted sleep in patients with treatment resistant schizophrenia (TRS) and by proxy lead to a reduction in psychotic symptoms and improvement in quality of life.

We are including treatment-resistant patients with schizophrenia other nonorganic and chronic psychoses and in addition meeting the criteria of a sleep or circadian disorder. Included patients will be block randomized to either 8-10 sessions of CBT-I (active treatment) with a specific focus on sleep or 8-10 sessions of regularCBT with a specific focus on patients' psychopathology (treatment as usual) approx.1 session/week.

After 12 weeks the full battery of assessments will be repeated forboth groups. Primary analyses will be to identify group-difference in changes using repeated measure ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ICD-10 schizophrenia (DF20), chronic paranoid psychosis (DF22), schizo-affective disorder (DF25) or other non-organic psychosis (DF28-DF29)
* Treatment resistance according to TRRIP criteria
* Sleeping difficulties (minimum duration 3 months)
* ISI score >14
* Stable psychopharmacological treatment the last month
* Only legal competent patient can participant

Exclusion Criteria:

* Psychiatric admission last six months (more than 1 week or resulted in significant changes in psychopharmacological treatment)
* Substance abuse to a degree that will interfere with participation.
* Diagnoses of sleep apnea/CPAP use

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | Baseline, after 12-weeks and 24-weeks.
  Patient-entered questionnaire measuring sleep difficulties. Seven items. Range of score 0-28. Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Positive and negative syndrome scale (PANSS) | Baseline, after 12-weeks and 24-weeks.
  32-items clinician administered rating scale measuring psychopathology. Range of score 30-210. Higher scores indicate higher level of symptoms
WHO well being index | Baseline, after 12-weeks and 24-weeks.
  5-five items patient-entered questionnaire. Measuring quality of life. Range of score 0-100. Higher scores indicate better quality of life.
Global Assessment of Functioning (GAF) | Baseline, after 12-weeks and 24-weeks.
  Rating scale measuring level of functioning. Clinician administered. Range of score 0-100. Higher scores indicate higher level of functioning.
Functioning Assessment Short Test (FAST) | Baseline, after 12-weeks and 24-weeks.
  Clinician administered rating scale measuring level of functioning. Range of score 0-72. Higher scores indicate lower level of functioning.
Personal and Social Performance scale | Baseline, after 12-weeks and 24-weeks.
  Semi-structured interview. Measuring level of functioning. Range of score 0-100. Higher scores indicate higher level of functioning.
Process of recovery questionnaire (QPR) | Baseline, after 12-weeks and 24-weeks.
  Questionnaire. Range 0-60. Higher scores indicate better outcome.
Sleep onset latency (PSG) | Baseline and after 12-weeks.
  Time until sleep verified by polysomnography. Measured in minutes. Increasing number is associated with poorer sleep.
Sleep efficiency (PSG) | Baseline and after 12-weeks.
  Time with verified sleep divided by Time spent in bed and multiplied by 100. Measured by polysomnography. Higher percentage is associated with better sleep quality.
Wake after sleep onset, number of awakenings (PSG) | Baseline and after 12-weeks.
  Number of wake periods after initial onset of sleep. Measured in number of awakenings . Higher number is associated with poorer sleep quality.
Wake after sleep onset, duration of wake periods (PSG) | Baseline and after 12-weeks.
  Duration of wake periods after initial onset of sleep. Measured in minutes of duration. Longer duration is associated with poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Nielsen, MD, Study Director — Psykiatrisk Center Glostrup
Locations (1):
- Mental Health Centre Glostrup, Glostrup, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman D, Waite F, Startup H, Myers E, Lister R, McInerney J, Harvey AG, Geddes J, Zaiwalla Z, Luengo-Fernandez R, Foster R, Clifton L, Yu LM. Efficacy of cognitive behavioural therapy for sleep improvement in patients with persistent delusions and hallucinations (BEST): a prospective, assessor-blind, randomised controlled pilot trial. Lancet Psychiatry. 2015 Nov;2(11):975-83. doi: 10.1016/S2215-0366(15)00314-4. Epub 2015 Sep 9. PMID 26363701
- [Background] Kaskie RE, Graziano B, Ferrarelli F. Schizophrenia and sleep disorders: links, risks, and management challenges. Nat Sci Sleep. 2017 Sep 21;9:227-239. doi: 10.2147/NSS.S121076. eCollection 2017. PMID 29033618
- [Background] Nucifora FC Jr, Woznica E, Lee BJ, Cascella N, Sawa A. Treatment resistant schizophrenia: Clinical, biological, and therapeutic perspectives. Neurobiol Dis. 2019 Nov;131:104257. doi: 10.1016/j.nbd.2018.08.016. Epub 2018 Aug 29. PMID 30170114
- [Background] Reeve S, Sheaves B, Freeman D. Sleep Disorders in Early Psychosis: Incidence, Severity, and Association With Clinical Symptoms. Schizophr Bull. 2019 Mar 7;45(2):287-295. doi: 10.1093/schbul/sby129. PMID 30202909
- [Background] Robertson I, Cheung A, Fan X. Insomnia in patients with schizophrenia: current understanding and treatment options. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Jun 8;92:235-242. doi: 10.1016/j.pnpbp.2019.01.016. Epub 2019 Jan 29. PMID 30707986